CLINICAL TRIAL: NCT01590862
Title: ON/OFF Stimulation and Reward Motivation in Patients With Deep Brain Stimulators
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Massachusetts General Hospital (Other)
Responsible Party: Principal Investigator, Darin Dougherty, MD, Associate Professor of Psychiatry, Massachusetts General Hospital
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 2011P002821
Record Dates: First submitted 2012-04-27; First posted 2012-05-03 (Estimated); Last update posted 2024-01-12 (Actual); Status verified 2024-01

CONDITIONS: Obsessive Compulsive Disorder; Major Depressive Disorder; Epilepsy
MeSH Terms: conditions — Obsessive-Compulsive Disorder; Depressive Disorder, Major; Epilepsy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (2):
- Deep Brain Stimulation On (Active Comparator): We will assess Reward Motivation behavior with Deep Brain Stimulation on.
  Interventions: Device: Deep Brain Stimulator
- Deep Brain Stimulation Off (No Intervention): We will assess Reward Motivation behavior with Deep Brain Stimulation off.

INTERVENTIONS:
Device: Deep Brain Stimulator — Medtronic Deep Brain Stimulation device turned on and off
  Arms: Deep Brain Stimulation On

SUMMARY:
We propose to study approach/avoidance behavior as measured by the Approach Avoidance task in 20 epilepsy patients undergoing implementation of depth electrodes for seizure monitoring in the Epilepsy Monitoring Unit at MGH. We will also study the effects of VC/VS electrical stimulation on approach-avoidance conflict in 20 adult patients who have undergone DBS implantation for severe MDD and/or OCD. There are 100-200 patients in the world with DBS electrodes in the VC/VS, and our research team cares for more than any other institution. Both participant groups will be assessed with respect to reward-aversion decision conflict using the task. The task will be performed with concurrent EEG recordings in DBS patients, and with continuous recording through our invasive neurophysiology rig in EMU subjects.

DETAILED DESCRIPTION:
DBS Patients:

The study will take place at a clinical office in the Charlestown Navy Yard (CNY), and will consist of one 8 hour visit with an optional second 8 hour visit, for a potential total of 16 hours. Study staff will schedule a convenient time for patients to arrive, or the research visit may be paired with a regularly scheduled DBS programming visit. A member of the Division of Neurotherapeutics authorized to manipulate DBS programming will turn the device on and off during the study. The subject's therapeutic parameters of the DBS system will not be changed. The subject will be asked to complete several questionnaires Beck Depression Inventory-II, Quick Inventory of Depressive Symptomatology, Snaith Hamilton Pleasure Scale, Mood and Anxiety Symptoms Questionnaire, and the Cognitive-Behavioral Avoidance Scale.

Following these questionnaires, a member of the study staff will teach the subjects to perform a modified version of the Approach-Avoidance task (adapted from Aupperle et al., in press and Amemori & Graybiel, 2012). Participants will be given a choice between a monetary reward (approach condition) plus an aversive stimulus (mild electric current further described below) or no monetary reward plus no aversive stimulus (avoid condition). Two partially filled rectangles (one red and one blue) will indicate the relative amount of potential punishment and reward. Subjects will use a joystick to direct a circle from a center fixation point to select either a plus sign associated with the approach condition or a square associated with the avoid condition. Subjects therefore control the outcome of each trial and whether or not they receive any aversive stimuli. After the task, participants will complete the AAC Task: Post-Questionnaire (adapted from Aupperle et al.)

The aversive stimulus is delivered in the form of a mild half second stimulation to the ankle at a level of their choice that is uncomfortable but not painful. This electrical current is produced by the Digitimer DS8R Constant Current Stimulator (Digitimer North America, LLC. Ft. Lauderdale, FL). Its previous model DS71 has been safely implemented in studies with previously MGH-approved IRB's (Milad et al., 2013). Patients will complete the task with DBS ON and DBS OFF. Because we are not changing the therapeutic parameters of stimulation, subjects should not experience any changes during the ON condition. Should any discomfort arise in the OFF condition, the subject will be able to terminate the study and return to the ON condition immediately.

Electroencephalography recordings (EEG) will be collected at 1450 Hz throughout the task in the ON and OFF conditions, using a Brain Research Products 96-channel active EEG system. Before each task run, we will also collect eyes-open and eyes-closed resting data, aiming for at least 1 min of data free from any eyeblink, muscle, or other artifact. All recordings will take place in a sound-isolated room, with careful scalp and electrode preparation to keep impedances under 5 kΏ. Ground/references will be in the midline to minimize hemispheric effects, and simultaneous EOG will permit blink/eyeroll artifact correction. The EEG system includes a camera, tracking devices, and software optimized for registration. All electrode positions will be digitized and referenced to subjects' pre-operative MRIs, enabling source-localized analysis.

Epilepsy Patients:

We will administer the same Ap-Av task in 20 epilepsy patients undergoing implantation of depth electrodes for seizure monitoring in the Epilepsy Monitoring Unit at MGH. Epilepsy unit experiments will involve both recording and stimulation. Recordings with the Ap-Av task will be collected throughout the clinical stay. At the end of the stay, there are 1-2 days when the patient resumes anti-seizure medications and the risk of a stimulation induced seizure is low. On those days, we will attempt to modify task behavior through stimulation. Based on our prior experience, we expect to test 1-2 stimulation targets per patient. In the first 10 patients, we will seek to replicate results that pregenual ACC stimulation leads to increased avoidance. On a randomly selected 50% of trials (interleaved so that patients are blind to stimulation), we will bilaterally stimulate the pregenual ACC (single bipolar pair per hemisphere) at 130 Hz and 2 mA, for 600 ms during cue presentation. In the subsequent 10 patients, we will attempt to extend the result that dACC theta power predicts approach behavior. When theta power rises above a set threshold (determined during the recording-only days), we will again stimulate the pACC.

For patients who have been implanted with clinical intracranial electrodes (whether or not they have also been implanted with research electrodes), additional scalp electrodes may be used. Usually, some electrodes are placed on the scalp for clinical purposes (as decided on by the clinical team). Patients receiving depth electrodes, for example, usually receive a standard set of scalp electrodes as well. However, if the clinical team decides that only a very small number of electrodes are needed for their purposes we may supplement this further with less than 10 additional electrodes. For this purpose, routinely-used clinical scalp electrodes (including EOG and EMG) will be employed. The exact number and placement will be constrained by clinical parameters. Specifically, regions close to any wound will be avoided to minimize the risk of infection. Also, as the clinical recording systems have limited numbers of channels, additional recording electrodes will be limited to what channels are available. In cases where a full set of scalp electrodes are used, the amount of time they are on the patient's head will be limited to approximately one day to decrease the risk of infection. This additional recording will be done one day before the scheduled date for removal of the intracranial electrodes.

ELIGIBILITY:
DBS Patients:

Inclusion Criteria:

• Deep brain stimulator implantation performed at least three months prior to study

Exclusion Criteria:

* Subjects unable to visualize stimulus objects with correction
* Dementia or other known cognitive deficit

Psychiatric Patients:

Inclusion Criteria:

* Right-handed (as determined by the Handedness Inventory; Oldfield,1971)
* Normal or corrected-to normal vision and hearing
* Current diagnosis of MDD or OCD

Exclusion Criteria for Patients:

* Clinical history of bipolar disorder
* Current or past psychotic disorder
* Gross structural brain damage
* Cognitive impairment that would affect a participant's ability to give informed consent
* Current substance abuse, or abuse within the past 3 months
* Clinical history of severe personality disorder
* Imminent risk of suicide or an inability to control suicide attempts
* Evidence of dementia or other significant cognitive impairment on neuropsychological evaluation

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2021-01-23 (Actual); Primary Completion 2025-03-31 (Estimated); Study Completion 2025-03-31 (Estimated)

PRIMARY OUTCOMES:
Approach Avoidance Task | Up to 8 hours for each visit
  The Approach Avoidance task is a computer task that assesses approach avoidance behavior. We will assess whether stimulation of the Ventral Capsule/Ventral Striatum has an effect on behavior by executing this task with the DBS system on and off.

CONTACTS AND LOCATIONS:
Overall Officials: Darin Dougherty, MD, Principal Investigator — Massachusetts General Hospital
Locations (2):
- United States (2):
  - Massachusetts General Hospital, Boston, Massachusetts
  - Massachusetts General Hospital, Charlestown, Massachusetts